CLINICAL TRIAL: NCT06679153
Title: A Randomized, Double-masked, Active-controlled, Multi-center Phase 2 Clinical Study Evaluating the Efficacy and Safety of 0.5% and 1.0% VVN461 Ophthalmic Solution in Patients With Noninfectious Anterior Uveitis
Brief Title: A Phase 2 Study of VVN461 Ophthalmic Solution for Noninfectious Anterior Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VivaVision Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVN461-CCS-201
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Anterior Uveitis
MeSH Terms: conditions — Uveitis, Anterior | interventions — prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VVN461, 1.0% (Experimental): VVN461 Ophthalmic Solution, 1.0%
  Interventions: Drug: VVN461 Ophthalmic Solution 1.0%
- VVN461, 0.5% (Experimental): VVN461 Ophthalmic Solution, 0.5%
  Interventions: Drug: VVN461 Ophthalmic Solution 0.5%
- Prednisolone acetate, 1% (Placebo Comparator): Prednisolone acetate Ophthalmic Solution, 1%
  Interventions: Drug: Prednisolone acetate

INTERVENTIONS:
Drug: VVN461 Ophthalmic Solution 1.0% — VVN461 Ophthalmic Solution, 1.0%, for up to 28 days
  Arms: VVN461, 1.0%
Drug: VVN461 Ophthalmic Solution 0.5% — VVN461 Ophthalmic Solution, 0.5%, for up to 28 days
  Arms: VVN461, 0.5%
Drug: Prednisolone acetate — Prednisolone acetate, 1%, for up to 28 days
  Other Names: Pred Forte
  Arms: Prednisolone acetate, 1%

SUMMARY:
This is a multicenter, double-masked, randomized, active-controlled, parallel-comparison study conducted at sites in the China in subjects with Noninfectious Anterior Uveitis

DETAILED DESCRIPTION:
In this study, subjects who meet the inclusion/exclusion criteria will be randomized to receive one of the three treatments prednisolone acetate during the Screening/Baseline Visit (Day-2 to Day 1). Starting from Visit 1 (Day 1), subjects will be administered one drop of the investigational product in the study eye in following dose regimens: 6 times per day (Q2h, 2 hours apart) for 7 days; 4 times per day (QID) for 7 days；2 times per day (BID) for 7 days；once a day (QD) for 7 days. Subjects will return to clinic for study assessments on Day 3 (Visit 2), Day 7 (Visit 3), Day 14 (Visit 4), Day 21 (Visit 5) and Day 28 (Visit 6, end of study) or early withdrawal/termination visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years at the time providing signed informed consent
* At least 1 eye diagnosed with noninfectious anterior uveitis at the time of screening
* Willing and able to comply with study requirements and visit schedule

Exclusion Criteria:

* Diagnosis of intermediate uveitis, posterior uveitis or panuveitis in either eye at the time of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
ACC score of ≥2 grade from baseline at Day 14 | Day 14
  Proportion of subjects with improvement in ACC score of ≥2 grade from baseline at Day 14

SECONDARY OUTCOMES:
ACC score of 0 | Baseline to Day 28
  Proportion of subjects with an ACC score of 0 at any visit

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China